CLINICAL TRIAL: NCT03349073
Title: An Extension Study of T-1101 (Tosylate) Administered Orally to Patients With Advanced Refractory Solid Tumors
Brief Title: An Extension Study for T-1101 (Tosylate) to Treat Advanced Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taivex Therapeutics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAI-002
Record Dates: First submitted 2017-11-17; First posted 2017-11-21 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Advanced Refractory Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T-1101 (Tosylate) (Experimental)
  Interventions: Drug: T-1101 (Tosylate)

INTERVENTIONS:
Drug: T-1101 (Tosylate) — T-1101 (Tosylate) powder in bottle

SUMMARY:
T-1101 is a novel anti-cancer agent being developed by Taivex Therapeutics Corporation, and is being studied in a phase I dose escalation trial, protocol TAI-001. That trial's primary aim is to study the safety and tolerability of T-1101 (Tosylate) in subjects with advanced refractory solid tumors, and provides for a maximum of 2 cycles of treatment. At the end of 2 cycles of treatment, it is likely that some patients will be continuing to receive clinical benefit from T-1101 (Tosylate). The intention of this program is to enable these patients to continue to receive T-1101 (Tosylate) at the discretion of the principal investigators and Taivex Therapeutics Corporation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced malignancy who are receiving T-1101 (Tosylate) in a previous Taivex Therapeutics Corp. sponsored study that has reached its endpoint, and who are, in the opinion of the investigator and/or sponsor, expected to continue to have an overall positive benefit/risk from continuing treatment.
2. Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation, including the 30 days period after last study drug dosing.
3. Women of childbearing potential who have a negative pregnancy test within 7 days of the first dose of T-1101 (Tosylate) in this long term extension trial.
4. Patients who have completed the End of Study assessments in their originating study. Every effort should be made to conduct the End of Study visit such that the patient does not have any interruption in T-1101 (Tosylate) dosing.
5. Signed and dated informed consent document indicating that the patient has been informed of all the pertinent aspects of the trial prior to enrollment.
6. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Any medical condition that, in the opinion of the investigator and/or sponsor, could jeopardize the safety of the patient.
2. Hypertension that cannot be controlled by medications (>150/100 mmHg despite optimal medical therapy).
3. Progressive or untreated metastatic brain or meningeal tumors.
4. Pregnancy or breastfeeding. Male patients must be surgically sterile or must agree to use effective contraception during the period of therapy. Female patients must be surgically sterile or be postmenopausal, or must agree to the use of highly effective contraception during the period of therapy. Highly effective method of birth control is defined as one that results in a low failure rate (i.e. less than 1 percent per year) when used consistently and correctly, such as implants, injectables, combined oral contraceptives, intra-uterine devices (IUDs), sexual abstinence, or a vasectomized partner.
5. Substance abuse, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

PRIMARY OUTCOMES:
Clinical Tumor Response of T-1101 (Tosylate) in Participants with Advanced Cancers Categorization of response based on RECIST 1.1. | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (4):
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - National Cheng Kung University (NCKU) Hospital, Tainan
  - Taipei Medical University Hospital, Taipei
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No